CLINICAL TRIAL: NCT00349102
Title: Evaluation of the Interest of Breath Holding for the Prevention of Radiation Pneumonitis Following Conformal Radiation Therapy
Brief Title: Prevention of Radiation Pneumonitis After Three-dimensional Conformal Radiation Therapy (3D-CRT) in Patients With Non-small-cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GATING 2006; ET2005-052
Record Dates: First submitted 2006-07-05; First posted 2006-07-06 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Carcinoma, Non-small-cell Lung
Keywords: Non-small-cell lung cancer; Breath-hold; Radiation pneumonitis; Serum cytokines; LENT-SOMA scale; Non-metastatic non-small-cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Radiation Pneumonitis | interventions — Breath Holding

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Free breathing during conformal radiation
  Interventions: Radiation: Free breathing
- B (Experimental): Breath holding during conformal radiation
  Interventions: Radiation: Breath holding

INTERVENTIONS:
Radiation: Free breathing — Free breathing during conformal radiation
  Other Names: Conformal radiation; Lung cancer
  Arms: A
Radiation: Breath holding — Breath holding during conformal radiation
  Other Names: Conformal radiation; Lung cancer
  Arms: B

SUMMARY:
The purpose of this study is to evaluate the interest of breath holding for the prevention of radiation pneumonitis following conformal radiation therapy.

Eligible patients will be randomly assigned in a 2-arm trial to free breathing or breath holding during conformal radiation.

The primary objective of the study is to establish the efficacy of breath holding, compared to free breathing, in the prevention of early pulmonary toxicity following conformal radiation.

Several departments of radiotherapy, many pneumology units and two basic and applied research laboratories take part in this multicentric study.

The number of patients required to demonstrate a reduction in radiation pneumonitis from 45 % to 22.5 %, assuming an alpha risk of 5% in a two-sided test and 95% power, is 240 (120 per arm). With a planned accrual of 7 patients per month, it is estimated that the inclusion period should be approximately 3 years.

DETAILED DESCRIPTION:
The secondary objectives are:

* Validation of the Lent-Soma toxicity scale by comparison to the RTOG scale,
* Response rate at different times: week 6-8, 1 year and 2 years after the end of irradiation,
* Progression-free survival rate at 1 year and 2 years after the end of irradiation
* Confirmation of the predictive value of serum cytokine levels (IL-6 and IL-10) during irradiation for the occurrence of early radiation toxicity, and analysis of the correlation between these serum levels at inclusion and the expression polymorphism of candidate genes.

ELIGIBILITY:
Inclusion Criteria:

* Non-metastatic cytologically or histologically proven non-small-cell lung cancer (NSCLC)
* Operated NSCLC patients requiring post-surgical irradiation or non-operated NSCLC patients requiring curative irradiation
* Conformational thoracic radiotherapy with curative intent
* Age >= 18
* Complete functional respiratory evaluation (FRE) performed less than 2 months before inclusion, demonstrating a maximum expiratory flow-volume/second > 1 l (in case surgery, the FRE must have been realized in the post-surgery period)
* Thoracic CT-scan performed less than 2 months before inclusion for non-operated patient
* PET-scan performed less than 2 months before inclusion for non-operated patient
* Performance status (PS) ECOG <= 1
* Possible training on breath holding technique
* Female patients of childbearing potential: effective method of contraception necessary
* Mandatory affiliation with a social security system
* Written, signed, informed consent

Exclusion Criteria:

* Small-cell lung cancer
* Metastatic disease
* Infiltrating pulmonary disease
* Previous thoracic irradiation
* Indication of irradiation with palliative intent
* Previous or concurrent primary malignancies at other sites (except basocellular skin cancer or cervical cancer in situ or complete remission for more than 5 years)
* Life expectancy < 6 months
* Patient understanding incompatible with the breath-hold technique (patients with major presbycusis are not eligible)
* Pregnant or lactating woman
* Patient included in another clinical trial
* Follow-up difficult
* Patient deprived of freedom

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2006-07 (Actual); Primary Completion 2012-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Clinical, functional and radiological evaluations at 6-8 weeks and 10-12 weeks after the end of irradiation | 6-8 and 10-12 weeks after the end of irradiation

SECONDARY OUTCOMES:
RTOG and LENT-SOMA scores at 6-8 weeks and 10-12 weeks after the end of irradiation, response rates at 6-8 weeks, 1 year and 2 years after irradiation | 6-8 and 10-12 weeks after the end of irradiation

CONTACTS AND LOCATIONS:
Overall Officials: Line CLAUDE, MD, Principal Investigator — Centre Leon Berard, Lyon
Locations (7):
- France (7):
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Institut Curie, Paris
  - Hôpital de la Pitié Salpêtrière, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Centre Catalan d'Oncologie, Perpignan
  - Centre René Gauducheau, Saint-Herblain

REFERENCES:
- [Background] Arpin D, Perol D, Blay JY, Falchero L, Claude L, Vuillermoz-Blas S, Martel-Lafay I, Ginestet C, Alberti L, Nosov D, Etienne-Mastroianni B, Cottin V, Perol M, Guerin JC, Cordier JF, Carrie C. Early variations of circulating interleukin-6 and interleukin-10 levels during thoracic radiotherapy are predictive for radiation pneumonitis. J Clin Oncol. 2005 Dec 1;23(34):8748-56. doi: 10.1200/JCO.2005.01.7145. PMID 16314635
- [Background] Claude L, Perol D, Ginestet C, Falchero L, Arpin D, Vincent M, Martel I, Hominal S, Cordier JF, Carrie C. A prospective study on radiation pneumonitis following conformal radiation therapy in non-small-cell lung cancer: clinical and dosimetric factors analysis. Radiother Oncol. 2004 May;71(2):175-81. doi: 10.1016/j.radonc.2004.02.005. PMID 15110451
- [Result] L. Falchero, D. Perol, D. Arpin, M. Vincent, M. Perol, JF. Cordier, D. Boutry, I. Martel-Lafay, C. Carrie.- Conséquences fonctionnelles de la radiothérapie thoracique conformationnelle (r3d) et facteurs prédictifs de pneumopathie radique aiguë (PRA) chez des patients atteints de cancer bronchique non à petites cellules (CNPC). Rev. Mal. Resp., 2001 ; 18 (suppl) : 1S102